CLINICAL TRIAL: NCT06733675
Title: A Phase 1, Open-label Study to Evaluate the Safety and to Characterize the Pharmacokinetics of a Fixed-Dose Combination Formulation of Ceftibuten-Ledaborbactam Etzadroxil
Brief Title: Safety and PK of Ceftibuten-ledaborbactam Etzadroxil Fixed-dose Combination
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VNRX-7145-106
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteer; Pharmacokinetics; Safety; Drug-Drug Interaction (DDI); FDC
Keywords: Healthy Volunteers; Ceftibuten; Ledaborbactam etzadroxil
MeSH Terms: interventions — Ceftibuten; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 (Experimental): Part 1 will enroll at least 16 participants who will receive a single oral dose of ceftibuten and ledaborbactam etzadroxil following a 10-hour fast on 3 occasions in a fixed sequence: (a) Ceftibuten and ledaborbactam etzadroxil as separate capsules; (b) Ceftibuten-ledaborbactam etzadroxil as fixed-dose combination capsules; (c) Ceftibuten-ledaborbactam etzadroxil as fixed-dose combination capsules after 5 days of esomeprazole orally once daily
  Interventions: Drug: Ledaborbactam etzadroxil; Drug: Ceftibuten; Drug: Ceftibuten-ledaborbactam etzadroxil; Drug: Esomeprazole
- Part 2 Group 1 (Experimental): Part 2 Group 1 will enroll 10 participants. Each will receive oral doses of Ceftibuten-ledaborbactam etzadroxil as fixed-dose capsules for 7 days (Fasted Group)
  Interventions: Drug: Ceftibuten-ledaborbactam etzadroxil
- Part 2 Group 2 (Experimental): Part 2 Group 2 will enroll 10 participants. Each will receive oral doses of Ceftibuten-ledaborbactam etzadroxil as fixed-dose capsules for 7 days (Fed Group)
  Interventions: Drug: Ceftibuten-ledaborbactam etzadroxil
- Part 2 Group 3 (Experimental): Part 2 Group 3 will possibly enroll 10 participants. Following availability of PK and safety data from Groups 1 and 2, a determination will be made regarding whether or not Group 3 is needed and the dosing conditions that apply
  Interventions: Drug: Ceftibuten-ledaborbactam etzadroxil

INTERVENTIONS:
Drug: Ledaborbactam etzadroxil — capsules
  Arms: Part 1
Drug: Ceftibuten — capsules
  Arms: Part 1
Drug: Ceftibuten-ledaborbactam etzadroxil — Fixed Dose Combination (FDC)
Drug: Esomeprazole — 40 mg capsule
  Arms: Part 1

SUMMARY:
This is a Phase 1, open-label, two-part, study in approximately 46 healthy adult participants between 18 and 55 years of age (both inclusive) (at least 16 participants in Part 1 and up to 30 participants in Part 2). The study will be conducted at one clinical site in the United States. Participants in Part 1 and Part 2 may be conducted in parallel. The duration of an individual participation will be approximately 46 days for Part 1 and 43 days for Part 2. All participants will be screened within 28 days prior to dosing. They will be admitted to the clinical research unit (CRU) the day prior to dosing and will remain in the CRU until the end of the PK sample collection period. All participants will return to the clinic for follow-up assessments 7 days ± 1 day after the last dose of study intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female, between 18 and 55 years of age
* Body mass index ≥ 18 and ≤ 32 kg/m2
* Laboratory values meeting defined laboratory ranges
* Males or non-pregnant, non-lactating females

Exclusion Criteria:

* History of any hypersensitivity reaction following administration of a cephalosporin, penicillin, or other β-lactam antibacterial drug
* Any acute illness or surgery within the past 3 months determined by the investigator to be clinically relevant
* Positive alcohol, drug or tobacco use/test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Part 1 Plasma PK AUC0-∞ (ceftibuten, ledaborbactam, and ledaborbactam etzadroxil) | 0 - 48 hours on days 1, 4 and 11
  Area under the concentration time curve from time zero to infinity (AUC0-∞)
Part 1 Plasma PK Cmax (ceftibuten, ledaborbactam, and ledaborbactam etzadroxil) | 0 - 48 hours on days 1, 4 and 11
  Maximum observed concentration (Cmax)
Proportion of participants of Part 2 experiencing Treatment-emergent adverse events (TEAEs), Serious TEAEs, or TEAEs leading to discontinuation. | Day 1 thru Day 18 (+/-1)
  Participants experiencing Treatment-emergent adverse events (TEAEs), Serious TEAEs, or TEAEs leading to discontinuation.

SECONDARY OUTCOMES:
Proportion of participants of Part 1 experiencing Treatment-emergent adverse events (TEAEs), Serious TEAEs, or TEAEs leading to discontinuation. | Day 1 thru Day 18 (+/-1)
  Participants experiencing Treatment-emergent adverse events (TEAEs), Serious TEAEs, or TEAEs leading to discontinuation.
Part 2 Plasma PK AUC0-12h (ceftibuten, ledaborbactam, and ledaborbactam etzadroxil) | Day 1 and Day 7
  Area under the concentration time curve from time zero to 12h (AUC0-12h)
Part 2 Plasma PK Cmax (ceftibuten, ledaborbactam, and ledaborbactam etzadroxil) | Day 1 and Day 7
  Maximum observed concentration (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Hamed, MD, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (1):
- ICON, Clinical Research Phase I Unit, Lenexa, Kansas, United States